CLINICAL TRIAL: NCT01575678
Title: The Effect of Melatonin on Nocturnal Enuresis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EnuMel-11; 2011-004138-33 (EudraCT Number)
Record Dates: First submitted 2012-02-24; First posted 2012-04-11 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Nocturnal Enuresis
Keywords: enuresis; melatonin; circadian rhythm; children; blood pressure; urine production; activity; sleep
MeSH Terms: conditions — Nocturnal Enuresis; Enuresis; Motor Activity | interventions — Melatonin; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Active Comparator)
  Interventions: Drug: Melatonin
- Lactose (Placebo Comparator)
  Interventions: Drug: Lactose

INTERVENTIONS:
Drug: Melatonin — blinded capsule 2-4 mg/day, oral use, for 4 weeks
  Arms: Melatonin
Drug: Lactose — blinded capsule 1/day, oral use, for 4 weeks
  Arms: Lactose

SUMMARY:
Aim: To investigate the effect of melatonin in bedwetting.

DETAILED DESCRIPTION:
Design: Double blind randomized placebocontrolled trial using crossover.

ELIGIBILITY:
Inclusion Criteria:

* Monosymptomatic nocturnal enuresis
* Age 6-14 years
* Clinical examination normal
* ≥ 3 wet nights / week due to either nocturnal polyuria with normal bladder size or reduced functional bladder capacity with normal urine output

Exclusion Criteria:

* Constipation (by ROME III criteria)
* Day incontinence
* Overactive bladder (ICCS 2008 classification of symptoms)
* Current or past history of clinical or laboratory findings that can be related to diseases or - conditions (eg pregnancy) likely to change the parameters examined, especially diseases of the kidney and urinary tract, liver or endocrine disorder.
* Clinical signs of urinary tract infection
* Hypertension, blood pressure assessed by ambulatory measurement with blood pressure cuff
* Set treatment with one or more drugs

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
number of incontinence episodes | 10 weeks

SECONDARY OUTCOMES:
nocturnal blood pressure | 4 weeks
  Time frame:
  Week 1: Baseline. Week 5: Effect of 1st treatment arm. Week 6: Wash out. Week 10: Effect of 2nd treatment arm.
activity level | 4 weeks
  Time frame:
  Week 1: Baseline. Week 5: Effect of 1st treatment arm. Week 6: Wash out. Week 10: Effect of 2nd treatment arm.
bladder capacity | 4 weeks
  Time frame:
  Week 1: Baseline. Week 5: Effect of 1st treatment arm. Week 6: Wash out. Week 10: Effect of 2nd treatment arm.
nocturnal urine production | 4 weeks
  Time frame:
  Week 1: Baseline. Week 5: Effect of 1st treatment arm. Week 6: Wash out. Week 10: Effect of 2nd treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Rittig, MD, dr.med, Principal Investigator — Pediatric department, Aarhus Universityhospital, Denmark
Locations (1):
- Center of Child Incontinence, Pediatric department, Aarhus Universityhospital, Aarhus, Central Jutland, Denmark

REFERENCES:
- [Derived] Caldwell PH, Codarini M, Stewart F, Hahn D, Sureshkumar P. Alarm interventions for nocturnal enuresis in children. Cochrane Database Syst Rev. 2020 May 4;5(5):CD002911. doi: 10.1002/14651858.CD002911.pub3. PMID 32364251